CLINICAL TRIAL: NCT00503438
Title: Salto Talaris Anatomic Ankle Arthroplasty Outcomes Study
Brief Title: Ankle Joint Replacement Outcomes Study
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: T-STAS-001
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Post-Traumatic Arthritis; Septic Arthritis; Prior Ankle Fusion
Keywords: Arthritis; Osteoarthritis; Arthroplasty
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Arthritis, Infectious; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Salto Talaris Ankle: This is an Implant Registry of the approved Salto Talaris Ankle replacement device
  Interventions: Device: Salto Talaris Ankle

INTERVENTIONS:
Device: Salto Talaris Ankle — Salto Talaris Anatomic Ankle total joint prosthesis
  Other Names: Salto Talaris

SUMMARY:
This post market outcome study will look at the therapeutic results of the Salto Talaris Anatomic ankle prosthesis. The study population will consist of patients who will undergo an ankle arthroplasty procedure with a Salto Talaris ankle implant. An analysis will be conducted of the results, complications and revisions of this prosthesis based on the etiology for which the ankle arthroplasty was performed.

DETAILED DESCRIPTION:
This is a prospective, multi-center study that will capture the therapeutic results of the Salto Talaris Anatomic ankle prosthesis in the treatment of various ankle afflictions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that need an ankle joint replacement due to arthritis or failed prior fusion.
* Subjects who have failed standard conservative management of their ankle condition

Exclusion Criteria:

* Class IV or higher anesthetic risk
* Subjects who are not able to comply with the study procedures
* Known contraindications to joint replacement such as active infection, complete talar necrosis, insufficient quality of bone stock, ligament laxity, severe osteopenia, Charcot's arthropathy
* Unwilling to be followed for 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidates will be considered regardless of gender, race or ethnicity. The racial, gender and ethnic characteristics of the proposed patient population will reflect the demographics of the surrounding area.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2007-10-31 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Survivorship of Salto Talaris Ankle Implant | 10 years
  Count of participants without a failed ankle arthroplasty. Ankle arthroplasty will be considered as failed if the implant is revised or removed and the ankle fused.

SECONDARY OUTCOMES:
The American Orthopaedic Foot and Ankle Society (AOFAS) Score | Postoperatively at 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, 8 years, and 10 years
  AOFAS ankle evaluation form is a commonly used standardized assessment of foot and ankle function divided into three anatomic regions. The scale used for this study will be the Ankle-Hindfoot Scale that ranges from 0 to 100. A score of 100 points is the maximum for a patient presenting in excellent condition. The score decreases as pain, limited range of motion, daily activities, joint instability, and alignment are assessed.

OTHER OUTCOMES:
The Foot Function Index (FFI) | Postoperatively at 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, 8 years, and 10 years
  FFI is a specialized questionnaire answered by the patient. The questionnaire consists of three parts used to report clinical scores for the domains of activity limitation, function, and disability in patients with foot and ankle conditions. Each item rated on a 0 - 10 Likert scale. 0 represents no pain/disability, and 10 represents the worst pain imaginable/severe disability for each item. Higher scores indicate decreased function.
The Foot and Ankle Ability Measure (FAAM) | Postoperatively at 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, 8 years, and 10 years
  FAAM is a region-specific subject questionnaire to evaluate activities of daily living and sports. Answers for both scales are based on a Likert scale (4-0) of:
  4 - no difficulty 3 - slight difficulty 2 - moderate difficulty
  1 - extreme difficulty 0 - unable to do Patients are asked to answer each question with a single response that most clearly describes their condition. Patients are asked to mark not applicable (N/A) if the activity in question is limited by something other than their foot or ankle. A higher score indicates a higher level of physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Marks, Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - Foot and Ankle Center of South Texas, San Antonio, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Bonnin M, Judet T, Colombier JA, Buscayret F, Graveleau N, Piriou P. Midterm results of the Salto Total Ankle Prosthesis. Clin Orthop Relat Res. 2004 Jul;(424):6-18. doi: 10.1097/01.blo.0000132407.75881.a0. PMID 15241138
- [Background] Pyevich MT, Saltzman CL, Callaghan JJ, Alvine FG. Total ankle arthroplasty: a unique design. Two to twelve-year follow-up. J Bone Joint Surg Am. 1998 Oct;80(10):1410-20. PMID 9801209
- [Background] Wood PL, Deakin S. Total ankle replacement. The results in 200 ankles. J Bone Joint Surg Br. 2003 Apr;85(3):334-41. doi: 10.1302/0301-620x.85b3.13849. PMID 12729104